CLINICAL TRIAL: NCT02838953
Title: Diaphragmatic Mobility, Lung Hyperinflation and Effects of the Pulmonary Rehabilitation
Brief Title: Measurements of Diaphragmatic Mobility on COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Casa Di Cura Villa Serena SpA (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Clinicavillaserena
Record Dates: First submitted 2016-06-30; First posted 2016-07-20 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Ultrasonography; Respiratory Function Tests; Pulmonary Disease, Chronic Obstructive; Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- COPD patients (Experimental): COPD patients submitted to Pulmonary Rehabilitation according to the ATS/ERS statement.
  Interventions: Behavioral: Pulmonary Rehabilitation
- Control (No Intervention): Healthy individuals who will undergo the same COPD's evaluation protocol. As "healthy individuals" they will not participate to the Pulmonary Rehabilitation.

INTERVENTIONS:
Behavioral: Pulmonary Rehabilitation — Comprehensive intervention based on a thorough patient assessment followed by patient- tailored therapies that include, but are not limited to, exercise training, education, and behavior change, designed to improve the physical and psychological condition of people with chronic respiratory disease and to promote the long-term adherence to health-enhancing behaviors.
  Arms: COPD patients

SUMMARY:
To determine whether the COPD impairs the diaphragmatic mobility (DM), and verify improvements after an inpatient pulmonary rehabilitation (PR).

Ultrasonography on M-mode will assess the diaphragmatic mobility at rest breathing and at slow deep inspiration. Lung functions test, arterial blood gas analyses, six minute walk test will be also performed, on COPD patients and healthy subjects.

DETAILED DESCRIPTION:
The diaphragm pathophysiological changes occurring in chronic obstructive pulmonary disease (COPD) leads to functional inefficiency that strongly correlates to the loss of lung function. Muscle fiber shortening follows lung hyperinflation, resulting to a chronic mechanical disadvantage, which worsens in COPD exacerbations. The DM is mostly assessed with techniques that exposes the patient to risks. The ultrasonography on M-mode is easy to use, safe and measures directly the diaphragmatic dome displacement. The study aim to determine whether the COPD impairs the DM, and verify improvements after an inpatient PR.

Every COPD patient will comprise a standard evaluation that consists on lung function test, six minute walk test and arterial blood gas analyses, according to the American Thoracic Society/ European Respiratory Society (ATS/ERS) statements.

Within the second day of recovery the diaphragm mobility ultrasonographic (US) measurement will be assessed as follow: the patients positioned in a semi recumbent position (45 degrees).The US probe positioned between the anterior and mean axillary line, on the central right subcostal area, cranial and dorsal. The US wave perpendicularly on the posterior hemidiaphragm third (it is visualized as the hyperechogenic line behind the liver). The mobility assessed by M-mode while the patient breaths on tidal volume (rest breathing) and deep slow breathing (to Functional Residual Capacity).

The COPD patients classification and diagnosis will be according to the the Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria. Every patient, after the assessment will follow the PR as ATS/ERS statement on pulmonary rehabilitation. All patients will follow a routine of five days a week of physical exercise. The rehabilitation program consists on a 30 minutes calisthenic gymnastic once a day, 20 minutes of cycloergometer training activity twice a day. The aerobic cycloergometer training was set at 60%-70% of the maximum cardiac frequency determined by 220 minus the patients age. The patients will perform lower limbs strengths exercises, especially for the quadriceps and hamstring. During the in-hospital stay, the patients will receive regular prescribed medication and oxygen therapy according to the medical staff evaluation, which will be prescribed by the clinician in charge. The patients will also have respiratory physiotherapy, regarding the presence of lung secretion retain, and the need to expand unventilated areas.

The control group will be composed by healthy volunteers. The volunteers will be screened on their lung function. The subjects on the control group will be submitted to the same evaluation protocol regarding the spirometry and the M-mode ultrasonography.

Statistical analyses:

The qualitative description of the data will be made with percentages and frequency. The quantitative data described as means and standard deviation for the symmetrical distributions. The Kolmogorov-Smirnov test to determine distributions mean normality. A One-way analysis of variance (ANOVA) with repeated measurements and Bonferroni test will be used as post-hoc test to evaluate statistical significance. Within-group effect sizes will be calculated using the Cohen d coefficient interpretation. For all the study data, the P values lower than 0.05 will be consider significant. The investigators will use the Student T- test for independent sample for quantitative data and for comparisons between the COPD patients and control group and ANOVA to the comparisons within COPD group. The investigators will use Pearson's correlation test to measure the correlation between the diaphragmatic mobility and the lung functioning variables.

ELIGIBILITY:
Inclusion Criteria

* Clinical Diagnosis of Chronic Obstructive Pulmonary Disease (COPD)
* Informed consent signature

Exclusion Criteria:

* Subjects with Pneumothorax
* Subjects with Active hemoptyses
* Subjects with Acute heart failure
* Subjects with Systemic arterial hypertension
* Subjects with aortic aneurism
* Subjects who underwent Hepatic surgery
* Subjects who underwent Splenectomy surgery
* Subjects with Diaphragmatic paralysis Subjects with Neuromuscular diseases Subjects with Chronic orthopaedic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-03; Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic mobility | up to four weeks
  diaphragmatic craniocaudal displacement on centimeters (performed on M-mode, mobility measured on centimeters)

SECONDARY OUTCOMES:
Lung function (Spirometry) | up to four weeks
  measurements of Forced vital capacity (liters), Forced expiratory volume on the first second (liters), expiratory reserve volume (liters), Inspiratory capacity (liters), Vital capacity (liters), Inspiratory reserve volume (liters), Tidal Volume (liters),
Lung function (Body plethysmography) | up to four weeks
  Total Lung capacity (liters), Total gas volume (liters), Residual volume (liters).
Lung function (gas exchange) | up to four weeks
  measurements of carbon monoxide lung diffusion (DLCO) on milliliters/minute/millimeters of mercury.
Functional status (Six minute walking test) | up to four weeks
  measurement of the distance walked (in meters) on six minutes
measurements of arterial blood gas | up to four weeks
  arterial blood sampling to measure hydrogenic potential (Ph), arterial oxygen pressure (PaO2), arterial carbonic anhydride pressure (PaCO2), bicarbonate (HCO3). PaO2, PaCO2 and HCO3 are measured on millimeters of mercury (mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Camilo Corbellini, PhD, Principal Investigator — Respiratory Physiotherapist
Locations (1):
- Casa di Cura Villa Serena, Piossasco, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qaseem A, Wilt TJ, Weinberger SE, Hanania NA, Criner G, van der Molen T, Marciniuk DD, Denberg T, Schunemann H, Wedzicha W, MacDonald R, Shekelle P; American College of Physicians; American College of Chest Physicians; American Thoracic Society; European Respiratory Society. Diagnosis and management of stable chronic obstructive pulmonary disease: a clinical practice guideline update from the American College of Physicians, American College of Chest Physicians, American Thoracic Society, and European Respiratory Society. Ann Intern Med. 2011 Aug 2;155(3):179-91. doi: 10.7326/0003-4819-155-3-201108020-00008. PMID 21810710
- [Background] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Background] Cassart M, Pettiaux N, Gevenois PA, Paiva M, Estenne M. Effect of chronic hyperinflation on diaphragm length and surface area. Am J Respir Crit Care Med. 1997 Aug;156(2 Pt 1):504-8. doi: 10.1164/ajrccm.156.2.9612089. PMID 9279231
- [Background] Vestbo J, Hurd SS, Agusti AG, Jones PW, Vogelmeier C, Anzueto A, Barnes PJ, Fabbri LM, Martinez FJ, Nishimura M, Stockley RA, Sin DD, Rodriguez-Roisin R. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2013 Feb 15;187(4):347-65. doi: 10.1164/rccm.201204-0596PP. Epub 2012 Aug 9. PMID 22878278
- [Result] Boussuges A, Gole Y, Blanc P. Diaphragmatic motion studied by m-mode ultrasonography: methods, reproducibility, and normal values. Chest. 2009 Feb;135(2):391-400. doi: 10.1378/chest.08-1541. Epub 2008 Nov 18. PMID 19017880
- [Derived] Corbellini C, Boussuges A, Villafane JH, Zocchi L. Diaphragmatic Mobility Loss in Subjects With Moderate to Very Severe COPD May Improve After In-Patient Pulmonary Rehabilitation. Respir Care. 2018 Oct;63(10):1271-1280. doi: 10.4187/respcare.06101. Epub 2018 Jul 31. PMID 30065081